CLINICAL TRIAL: NCT02420054
Title: Effects of Short Term Intermittent Fasting on Insulin Resistance in Type 2 Diabetes
Brief Title: Short Term Intermittent Fasting and Insulin Resistance
Acronym: IFAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Flemming Dela, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Intermittent Fasting
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Obesity
Keywords: intermittent fasting; alternate day fasting; diabetes mellitus; non-alcoholic fatty liver disease; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Obesity; Intermittent Fasting; Insulin Resistance | interventions — Flowering time control protein FCA, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent fasting (Active Comparator): Intermittent fasting conducted by a group of subjects with type 2 diabetes mellitus and an age- and BMI matched control group.
  Interventions: Behavioral: Intermittent fasting
- Time control (Active Comparator): A time control period.
  Interventions: Other: Time control

INTERVENTIONS:
Behavioral: Intermittent fasting — Alternate day fasting (ADF) (water permitted) for 3 weeks with double energy intake every other day. Followed by ADF for 3 weeks with ad libitum diet on eating days.
  Arms: Intermittent fasting
Other: Time control — Time control period with no change in eating habits.
  Arms: Time control

SUMMARY:
The purpose of the study is to determine the effect of intermittent fasting on insulin secretion and insulin sensitivity in skeletal muscle and fat distribution.

DETAILED DESCRIPTION:
Approximately 250.000 patients are diagnosed with type 2 diabetes (T2DM) in Denmark, and world-wide close to 350 million people suffer from diabetes. T2DM develops in genetically susceptible individuals as a result of excess energy intake and insufficient amount of daily physical activity. The pathophysiology encompasses a mismatch between the insulin secretory capacity and insulin sensitivity, predominantly manifested in skeletal muscle as insulin resistance. T2DM is associated with increased morbidity and mortality.

The disease is triggered by the individual lifestyle, and thereby the potential for prevention and reversal of the disease in its early years after diagnosis is quite large.

One potential way to improve glucose homeostasis is by intermittent fasting, also known as alternate day fasting. Intermittent fasting means switching between eating and fasting, and it is a variation of calorie restriction. Intermittent fasting has been studied in animals. Together with calorie restriction, intermittent fasting is the most efficient way to expand lifespan of many animal species without genetically altering them. A wide range of age related changes are delayed including beneficial effects on hypertension, degenerative brain disease, immune responses, DNA repair capacity and glucose homeostasis. Fat redistribution with fat translocating from between the organs and the liver to the subcutis.

Little is known about intermittent fasting in humans. In 2005 the investigators experimentally tested this concept in young healthy males and found that 15 days of alternating days with fast and food intake increased insulin sensitivity by 16% without any changes in body weight.

The explanation could be oscillations in cellular energy stores. Skeletal muscle contains approximately 80% of the stored glycogen alone by virtue of the muscle mass. The liver has a higher glycogen concentration, but it is much smaller. A single prolonged (>24 hrs) day of fasting may not decrease muscle glycogen, while the decrease in the liver is very fast. A muscle glycogen lowering effect of continued intermittent fasting would be expected, and experimentally indicated.

The intermittent fasting method may appeal to some patients, who do not exercise, and the need for testing this intervention in patients with type 2 diabetes is obvious.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-35
* Type 2 diabetes or metabolically healthy
* Diet or orally administered treatment for type 2 diabetes

Exclusion Criteria:

* Regular physical activity
* Other diseases than type 2 diabetes
* insulin treatment
* alcohol abuse

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Insulin Sensitivity after 20 days of intermittent fasting. | 46 days
  An euglycemic hyperinsulinemic clamp is performed at day 1 and repeated at day 23 after a control period with no change in the diet. Baseline insulin sensitivity is determined based on these two measurements. The euglycemic hyperinsulinemic clamp is repeated at day 46 after the intermittent fasting period (day 25-44) and two days (day 24 and 45) with a normal diet.
Change of insulin secretion | 46 days
  IVGTT performed at baseline, after intermittent fasting without weight loss and again after intermittent fasting with weight loss

SECONDARY OUTCOMES:
Glycogen Content in Skeletal Muscle after a Day of Eating and after a Day of Fasting | 46 days
  Analysis of glycogen content from muscle biopsies obtained after a day of fasting and after a day of eating during the intermittent fasting period.
Change from Baseline in Fat Content in the Liver and Visceral Fat after 20 Days of Intermittent Fasting | 23 days
  Fat content measured by magnetic resonance spectroscopy.
Insulin signalling cascade proteins | 46 days
  By Western blot determine any change in proteins relevant for insulin signalling and turnover of intramyocellular lipids.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, MD, DMSc, Principal Investigator — University of Copenhagen
Locations (1):
- Xlab, Department of Biomedical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ingersen A, Helset HR, Calov M, Chabanova E, Harreskov EG, Jensen C, Hansen CN, Prats C, Helge JW, Larsen S, Dela F. Metabolic effects of alternate-day fasting in males with obesity with or without type 2 diabetes. Front Physiol. 2022 Dec 1;13:1061063. doi: 10.3389/fphys.2022.1061063. eCollection 2022. PMID 36531168